CLINICAL TRIAL: NCT02801812
Title: An Observational Multicenter International Case-control Study for the Assessment of Nailfold Capillary Abnormalities in Patients with Systemic Lupus Erythematosus
Brief Title: Observational Multicenter Case-control Study to Assess Nailfold Capillary Abnormalities in Systemic Lupus Erythematosus
Status: Completed | Type: Observational
Sponsor: ASST Gaetano Pini-CTO (Other)
Collaborators: EULAR study group on microcirculation in rheumatic diseases (Unknown)
Responsible Party: Principal Investigator, Ingegnoli Francesca, MD, PhD, ASST Gaetano Pini-CTO
Other Study IDs: SG_MC/RD4
Record Dates: First submitted 2016-06-13; First posted 2016-06-16 (Estimated); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Systemic Lupus Erythematosus
Keywords: Nailfold Capillaroscopy
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — Microscopic Angioscopy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Systemic Lupus Erythematosus: patients ≥18 years diagnosed SLE upon classification according to 2012 SLICC criteria and disease onset ≥16 years.
  Interventions: Device: nailfold capillaroscopy
- Healthy controls: subjects ≥18 years fulfilling the definition proposed in the protocol.
  Interventions: Device: nailfold capillaroscopy

INTERVENTIONS:
Device: nailfold capillaroscopy — Detection by nailfold capillaroscopy of capillary abnormalities in patients with Systemic Lupus Erythematosus and comparison with healthy controls at enrolment

SUMMARY:
The purpose of this study is to investigate the role of nailfold capillaroscopy in the assessment of patients with Systemic Lupus Erythematosus (SLE).

Primary endpoint:

- To compare the frequency of major capillaroscopic abnormalities in patients with SLE and healthy controls.

Secondary endpoints:

* To compare the frequency of major capillaroscopic abnormalities in patients with active and non-active SLE / active SLE and healthy controls / non-active SLE and healthy controls.
* To study the association of different capillaroscopic parameters and the status of subjects (SLE / active SLE / non-active SLE / healthy controls).

DETAILED DESCRIPTION:
Background and rationale:

Nailfold capillaroscopy (NC) is a diagnostic investigation used in the routine clinical setting for the differential diagnosis of connective tissue diseases, such as Systemic Lupus Erythematosus (SLE). Among SLE clinical manifestations, vascular involvement is a common feature and a variable prevalence of NC abnormalities has been reported in SLE: typical NC changes, as well as non-specific variations as observed in healthy subjects.

At this very moment literature is interspersed with different descriptions of capillaroscopic features in SLE, and it has not been clearly defined the role of NC in SLE patients. It has been suggested that the presence of major capillary abnormalities may reflect the microvascular systemic involvement in SLE, and it may correlate to the disease activity.

Against this background, the EULAR study group on microcirculation in rheumatic diseases planned an international multicenter study.

Objective:

To investigate the role of NC abnormalities in the assessment of SLE patients.

Endpoints:

Primary endpoint:

-To compare the frequency of major capillary abnormalities in patients with SLE and healthy controls.

Secondary endpoints:

* To compare the frequency of major capillary abnormalities in patients with active and non-active SLE / active SLE and healthy controls / non-active SLE and healthy controls.
* To study the association of different capillary parameters and the status of subjects (SLE / active SLE / non-active SLE / healthy controls).

No. of subjects:

Total entered: 364 ; Cases (SLE): 182 ; Controls: 182.

Variables

NC assessment: presence of major capillary abnormalities; NC parameters/mm: number of capillaries, presence of hairpin, tortuous, crossed, bushy, ramified, enlarged, giant capillaries, microhemorrhages, architecture disorganization, visibility of the subpapillary venular plexus; presence of scleroderma patterns, normal patterns.

Clinical assessment: all subjects: date of birth, gender, race. SLE: age at disease onset, disease activity (SLEDAI-2000) and damage index (SLICC-DI), presence of antinuclear antibodies, anti-dsDNA, anti-Extractable Nuclear Antigen antibodies, lupus anticoagulant, anticardiolipin/beta2glycoprotein I antibodies, Raynaud's phenomenon, Hypertension, active smoke, diabetes mellitus, ongoing and cumulative dose steroid treatment, ongoing immunomodulatory/suppressive treatment.

Statistical methods For the primary endpoint and similar secondary endpoints, McNemar test (matching design) and a conditional odds ratio (OR). For other secondary endpoints, the Fisher's exact test and an OR, and a conditional logistic regression model (matching design) and non-conditional regression model and OR as appropriate.

ELIGIBILITY:
Inclusion Criteria:

* At time of enrollment all subjects must be 18 years or older and give written consent.
* Patients with SLE must fulfill the 2012 SLICC classification criteria.
* SLE onset must be over 16 years of age.
* Patients with SLE and secondary anti-phospholipid syndrome will be also enrolled.
* Healthy controls will be selected according to the definition proposed in the protocol

Exclusion Criteria:

* Subject refuses to sign and/or he/she is not able to understand the patient informed consent.
* Subjects with periungual traumatic lesions that may create artifacts (i.e. recent manicure, onychophagia, or gardening).
* SLE overlapping with other rheumatic diseases such as Systemic Sclerosis, Rheumatoid Arthritis, Mixed Connective Tissue Disease, Sjögren's Syndrome, Dermatomyositis, Polymyositis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients ≥18 years diagnosed with SLE upon classification according to 2012 SLICC criteria and disease onset ≥16 years.
Sampling Method: Non-Probability Sample
Enrollment: 364 (Actual)
Dates: Start 2016-01; Primary Completion 2018-12 (Actual); Study Completion 2019-02 (Actual)

PRIMARY OUTCOMES:
major capillary abnormalities | Day 1
  To compare the frequency of major capillary abnormalities in patients with SLE and healthy controls.

CONTACTS AND LOCATIONS:
Overall Officials: Francesca Ingegnoli, MD, Principal Investigator — ASST Gaetano Pini-CTO

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Petri M, Orbai AM, Alarcon GS, Gordon C, Merrill JT, Fortin PR, Bruce IN, Isenberg D, Wallace DJ, Nived O, Sturfelt G, Ramsey-Goldman R, Bae SC, Hanly JG, Sanchez-Guerrero J, Clarke A, Aranow C, Manzi S, Urowitz M, Gladman D, Kalunian K, Costner M, Werth VP, Zoma A, Bernatsky S, Ruiz-Irastorza G, Khamashta MA, Jacobsen S, Buyon JP, Maddison P, Dooley MA, van Vollenhoven RF, Ginzler E, Stoll T, Peschken C, Jorizzo JL, Callen JP, Lim SS, Fessler BJ, Inanc M, Kamen DL, Rahman A, Steinsson K, Franks AG Jr, Sigler L, Hameed S, Fang H, Pham N, Brey R, Weisman MH, McGwin G Jr, Magder LS. Derivation and validation of the Systemic Lupus International Collaborating Clinics classification criteria for systemic lupus erythematosus. Arthritis Rheum. 2012 Aug;64(8):2677-86. doi: 10.1002/art.34473. PMID 22553077
- [Background] Gladman DD, Ibanez D, Urowitz MB. Systemic lupus erythematosus disease activity index 2000. J Rheumatol. 2002 Feb;29(2):288-91. PMID 11838846
- [Derived] Ingegnoli F, Ughi N, Riccieri V, Stefanantoni K, Cracowski JL, Gutierrez M, Sulli A, Rodriguez-Reyna TS, Hame A, Makol A, Nuno-Nuno L, Nieto-Gonzalez JC, Kubo S, Michalska-Jakubus M, Sanchez Pernaute O, De Angelis R, Herrick AL, Melsens K, Cutolo M, Smith V; EULAR Study Group on Microcirculation in Rheumatic Diseases collaborators. Distribution of nailfold videocapillaroscopy parameters in systemic lupus erythematosus and their association with disease activity: an international blinded case-control analysis on behalf of the EULAR study group on microcirculation in rheumatic diseases. RMD Open. 2025 Sep 8;11(3):e005772. doi: 10.1136/rmdopen-2025-005772. PMID 40921627